CLINICAL TRIAL: NCT07348861
Title: A Phase II, Prospective, Single-Arm, Multicenter, Open-Label Study of Sacituzumab Tirumotecan in Combination With Iparomlimab and Tuvonralimab as Neoadjuvant Therapy for Locally Advanced Cervical Cancer
Brief Title: A Phase II Study of Neoadjuvant Sacituzumab Tirumotecan in Combination With Iparomlimab and Tuvonralimab in Locally Advanced Cervical Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zheng Min (Other)
Collaborators: Sichuan Kelun-Biotech Biopharmaceutical Co., Ltd. (Industry); Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Zheng Min, Profeesor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2025-751-01
Record Dates: First submitted 2026-01-08; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Cervical Cancer
Keywords: Locally advanced cervical cancer; cervical cancer stage IB3 (FIGO2018); cervical cancer stage IIA2 (FIGO2018); tumor size ≥ 4 cm cervical cancer stage IIIc1r (FIGO2018)
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Intervention Model Description: Sacituzumab tirumotecan, 5mg/kg iv. drip，Q2W Iparomlimab and Tuvonralimab, 3mg/kg iv.drip, Q2W
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sacituzumab tirumotecan plus Iparomlimab (Experimental)
  Interventions: Drug: Sacituzumab tirumotecan plus Iparomlimab

INTERVENTIONS:
Drug: Sacituzumab tirumotecan plus Iparomlimab — Sacituzumab tirumotecan 5mg/kg iv. drip,Q2W Iparomlimab and Tuvonralimab 3mg/kg iv.drip, Q2W

SUMMARY:
This is a phase II, prospective, single-arm, multicenter, open-label study to evaluate the efficacy and safety of sacituzumab tirumotecan in combination with iparomlimab and tuvonralimab as neoadjuvant therapy in patients with locally advanced cervical cancer

DETAILED DESCRIPTION:
The goal of this clinical trial is to learn if Sacituzumab tirumotecan plus Iparomlimab and Tuvonralimab works to treat locally advanced cervical cancer. It will also learn about the safety of the combination of these two drugs. The main questions it aims to answer are:

* Does Sacituzumab tirumotecan plus Iparomlimab and Tuvonralimab increase the rate of pathological complete response?
* What medical problems do participants have when treating Sacituzumab tirumotecan plus Iparomlimab and Tuvonralimab? Researchers will calculate the rate of pathological complete response and collect the adverse events to see the efficacy and safety of Sacituzumab tirumotecan plus Iparomlimab and Tuvonralimab in locally advanced cervical cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary participation in the clinical study; complete understanding, knowledge of this study and signing informed consent; willingness to follow and ability to complete all trial procedures;
2. Histopathology confirmed cervical scaly carcinoma, adenocarcinoma, and adenocarcinoma. If there are small cell carcinomas, neuroendocrine carcinomas, and sarcoma components, they cannot be grouped ;
3. Locally advanced cervical cancer, according to FIGO2018 stage, conforming to stage IIB/IIIc1r with IB3, IIA2, and tumor diameter ≥ 4 cm;
4. Has not previously received any other anti-tumor treatment ;
5. Age 18-65 years ;
6. The physical fitness score of the Eastern U.S. Oncology Cooperation Group (ECOG) was 0 to 1 score ;
7. Life expectancy exceeds 3 months ;
8. Organ function and hematopoietic function must meet the following requirements:

   Hemoglobin (HGB) ≥80g/L; Leukocyte count (WBC) ≥ 3×109/L; absolute neutrophil count (ANC) ≥ 1.5 × 109/L ; Platelet count (PLT) ≥80×109/L; Total cholugin (TBIL) ≤ 1.5 × normal value upper limit (ULN) ; aspartate transaminase AST) and aspartate transaminase (ALT) ≤ 2.5 × ULN ; If hepatic dysfunction is caused by tumor hepatic metastasis, AST and ALT ≤ 5 × ULN ; Serum creatinine (Cr) ≤ 1.5 × ULN; or creatinine clearance rate (CrCl) ≥ 50 mL/min; International standardized ratio (INR) or plasma coagulase prime time (PT) ≤ 1.5 × ULN.
9. Female subjects in childbearing age must agree to effective contraception measures within 5 months after signing a informed consent form, during the study period, and after the last administration of the drug ;
10. Subjects must agree to provide sufficient tumor tissue samples for PD-L1, TROP2 expression detection. This includes archived tumor samples (paraffin blocks or untainted sections in quantity that meet the testing requirements specified by this institute); without archived tumor tissue samples, subjects agree to undergo tumor lesion rebiometry.

Exclusion Criteria:

1. Research treatments that have begun to receive other anti-tumor treatments (including chemotherapy, molecular targeting therapy, radiotherapy, immunotherapy, monoclonal antibody therapy), or that have participated in other non-marketing drug clinical studies ;
2. Subjects known to have previously been allergic to macromolecular protein preparations / monoclonal antibodies, or known to be allergic to the composition of any experimental drug ;
3. pregnant or breastfeeding women ;
4. Those with active autoimmune diseases and who have received systematic treatment (such as corticosteroids or immunosuppressive drugs) within the past 2 years (such as, but not limited to: meningitis, enteritis, hepatitis, pituitary, vascular, nephritis, hyperthyroidism, hypothyroidism [inclusive for non-clinical symptomatic hypothyroidism or hypothyroidism due to chemotherapy]; those with vitiligo or who had complete remission of asthma in childhood and need no intervention in adulthood;)
5. Whole-body corticosteroid (dosage equivalent to or greater than 10 mg/day strong pine) or other immunosuppressive drug therapists were required within 14 days prior to group admission or during the study period ;
6. Individuals who received live vaccination within 4 weeks of treatment initiation ;
7. Those who have received anti-tumor vaccines, or those who have received anti-tumor therapies with systemic immunostimulatory effects ;
8. With serious medical conditions, such as severe infections, uncontrollable diabetes, cardiovascular disease (classified by the New York Heart Association as Class III or IV heart failure, cardiovascular obstruction above Class II, myocardial infarction within the past 6 months, unstable arrhythmia or unstable angina, cerebral infarction within 3 months, etc.) or pulmonary disease (history of interstitial pneumonia, obstructive pulmonary disease, and symptomatic Bronchospasm);
9. Hepatitis C virus deoxyribonucleic acid (HBV DNA) > 103 copies/ml positive for hepatitis C surface antigen (HBsAg) and/or hepatitis C core antibody (HBcAb), or hepatitis C virus antibody positive; syphilis positive;
10. Has a history of human immunodeficiency virus infection, or has other acquired, congenital immunodeficiency diseases ;
11. Those with an active tuberculosis infection history within 1 year prior to group admission ;
12. Patients with other malignancies within 5 years of group entry, except for any previously cured type of in situ carcinoma and cured skin basal-cell carcinoma or skin scaly carcinoma ;
13. Previously received exogenous hematopoietic stem cell or solid organ transplantation ;
14. Those with a history of gastrointestinal perforation or who underwent excessive surgical surgery (excluding baseline tumor biopsies) or who suffered severe trauma, active ulcers, intestinal perforation, intestinal obstruction, and unhealed fractures within the first 4 weeks of study treatment ;
15. Has a history of alcoholism, drug use or drug abuse within the past 1 year ;
16. Having a clear history of neurological or mental disorders, such as epilepsy, dementia, and dependence disorder;
17. Other severe, acute, or chronic diseases or laboratory abnormalities that may increase the risk of participation in studies and study drug use, or may interfere with the interpretation of study results ;
18. People with previous eye surface disorders, e.g.: dry eye disease, corneal inflammation, etc. conditions ;
19. The presence of a relative or absolute taboo condition for abdominal cervical cancer surgery ;
20. Researchers consider participants unsuitable for this study due to other reasons.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Rate of pathological complete response | From enrollment to the end of treatment at 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
ICMJE